CLINICAL TRIAL: NCT04285580
Title: An Evaluation of the 24-Hour Intraocular Pressure(IOP)-Lowering Effect of Bimatoprost Sustained-Release(SR) in Participants With Open-Angle Glaucoma(OAG) or Ocular Hypertension(OHT)
Brief Title: A Phase 3b Study Evaluating the 24-Hour Intraocular Pressure Lowering Effect of Bimatoprost SR in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1698-304-007
Expanded Access: NCT05338606 (No longer available)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimatoprost SR 10 μg (Experimental): Participants will receive Bimatoprost SR 10 μg implant in the study eye on Day 1 and standard of care treatment in the fellow eye for the duration of the study.
  Interventions: Drug: Bimatoprost SR
- LUMIGAN 0.01% (Other): Participants will receive topical LUMIGAN 0.01% in the study eye once daily starting evening Dose on Day 1 and standard of care treatment in the fellow eye for the duration of the study.
  Interventions: Drug: LUMIGAN

INTERVENTIONS:
Drug: Bimatoprost SR — Consists of 1 Bimatoprost SR administration in the study eye.
  Arms: Bimatoprost SR 10 μg
Drug: LUMIGAN — Treatment with LUMIGAN 0.01% begins on Day 1. The drop will be instilled once daily in the evening to the study eye throughout the duration of the study.
  Arms: LUMIGAN 0.01%

SUMMARY:
This study will evaluate the 24-hour intraocular pressure lowering effect and safety after a single administration of Bimatoprost SR in patients with Open-Angle Glaucoma or Ocular Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either OAG or OHT study eye, requiring IOP-lowering treatment
* Participant is currently a nonsmoker and has not smoked any nicotine-containing products within the previous 6 months

Exclusion Criteria:

* Current or anticipated enrollment in another investigational drug or device study
* Females who are pregnant, nursing, or planning a pregnancy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2022-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (6):
- United States (6):
  - Trinity Research Group /ID# 232749, Dothan, Alabama
  - The Eye Research Foundation /ID# 232694, Newport Beach, California
  - Coastal Research Associates /ID# 232798, Roswell, Georgia
  - James D Branch MD /ID# 232718, Winston-Salem, North Carolina
  - Scott and Christie and Associates /ID# 232747, Cranberry Township, Pennsylvania
  - Keystone Research LTD /ID# 232665, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Weinreb RN, Christie WC, Medeiros FA, Craven ER, Kim K, Nguyen A, Bejanian M, Wirta DL. Single Administration of Bimatoprost Implant: Effects on 24-Hour Intraocular Pressure and 1-Year Outcomes. Ophthalmol Glaucoma. 2023 Nov-Dec;6(6):599-608. doi: 10.1016/j.ogla.2023.06.007. Epub 2023 Jun 19. PMID 37343625

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost SR 10 μg | LUMIGAN 0.01%
Started | 31 | 6
Completed | 31 | 5
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who have received study intervention (ie, Bimatoprost SR administration or LUMIGAN 0.01%) with at least 1 postbaseline IOP assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost SR 10 μg | LUMIGAN 0.01% | Total
Number analyzed (Participants) | 31 | 6 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 2 | 12
  >=65 years | 21 | 4 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (11.81) | 70.2 (8.52) | 70.4 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 2 | 20
  Male | 13 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 28 | 6 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 22 | 4 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Hour 0 Intraocular Pressure (IOP) [Count of Participants; unit: Participants]
  <= 25 mmHg | 26 | 3 | 29
  > 25 mmHg | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time-Matched Intraocular Pressure (IOP) for Bimatoprost SR Treated Eyes
Description: IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost SR 10 μg | LUMIGAN 0.01%
Number analyzed (Participants) | 31 | 5
Millimeters of Mercury (mmHg)
  Diurnal/Wake Period Hour 08:00 | -3.7 (5.65) | -4.0 (5.27)
  Diurnal/Wake Period Hour 10:00 | -2.5 (4.46) | -3.2 (3.09)
  Diurnal/Wake Period Hour 12:00 | -2.9 (3.36) | -5.0 (2.72)
  Diurnal/Wake Period Hour 14:00 | -1.8 (4.31) | -4.4 (2.04)
  Diurnal/Wake Period Hour 16:00 | -3.3 (3.80) | -4.2 (3.01)
  Diurnal/Wake Period Hour 18:00 | -1.9 (4.59) | -4.2 (2.08)
  Diurnal/Wake Period Hour 20:00 | -2.6 (4.29) | -5.0 (2.03)
  Diurnal/Wake Period Hour 22:00 | -2.3 (3.66) | -2.1 (2.48)
  Nocturnal/Sleep Period Hour 00:00 | -1.7 (3.60) | -1.8 (4.28)
  Nocturnal/Sleep Period Hour 02:00 | -2.4 (4.04) | -3.2 (3.25)
  Nocturnal/Sleep Period Hour 04:00 | -2.1 (3.85) | -3.2 (1.30)
  Nocturnal/Sleep Period Hour 06:00 | -2.2 (4.42) | -5.0 (3.34)

2. Primary Outcome: Number of Patients Experiencing One or More Treatment Emergent Adverse Events (TEAEs)
Description: The number of patients who experienced one or more TEAEs
Time Frame: Up to 12 Months
Population: All participants who have received study intervention (ie, Bimatoprost SR administration or LUMIGAN 0.01%)
Measure: Count of Participants; unit: Participants
Arm/Group | Bimatoprost SR 10 μg | LUMIGAN 0.01%
Number analyzed (Participants) | 31 | 6
Participants | 12 | 4

3. Secondary Outcome: Change From Baseline in Range of Intraocular Pressure (IOP) for Bimatoprost SR-treated Eyes
Description: IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening. The range of IOP is calculated as maximum value minus minimum value per participant for each corresponding period with the smaller values showing less fluctuation of IOP.
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost SR 10 μg | LUMIGAN 0.01%
Number analyzed (Participants) | 31 | 5
Millimeters of Mercury (mmHg) | -1.6 (2.98) | 0.7 (3.90)

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Bimatoprost SR 10 μg | LUMIGAN 0.01%
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/6
Other Adverse Events (participants affected / at risk) | 20/31 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimatoprost SR 10 μg (N=31) | LUMIGAN 0.01% (N=6)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimatoprost SR 10 μg (N=31) | LUMIGAN 0.01% (N=6)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 2 (3) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 3 (3) | 0 (0)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 11 (18) | 4 (8)
DRY EYE (Eye disorders) | 2 (3) | 0 (0)
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 2 (2) | 0 (0)
PUNCTATE KERATITIS (Eye disorders) | 2 (6) | 0 (0)
VISUAL FIELD DEFECT (Eye disorders) | 3 (4) | 0 (0)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 7 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT04285580/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT04285580/SAP_001.pdf